CLINICAL TRIAL: NCT00699283
Title: An International, Double-blind, Randomized, Multi-center, Parallel Group, Historical-control Conversion to Monotherapy Study to Evaluate the Efficacy and Safety of Brivaracetam in Subjects (≥ 16 to 75 Years Old) With Partial Onset Seizures With or Without Secondary Generalization.
Brief Title: A Double-blind, Randomized Conversion to Monotherapy Study to Evaluate the Efficacy and Safety of Brivaracetam in Subjects (≥ 16 to 75 Years Old) With Partial Onset Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: An interim analysis revealed the study was unlikely to attain a positive outcome for the efficacy analysis. No safety concerns were detected
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01306; RPCE07F1216; 2008-000145-58 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Monotherapy; Partial Onset Seizures; Adults and Adolescents
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brivaracetam (BRV) 1 (Experimental): 50 mg daily
  Interventions: Drug: Brivaracetam
- Brivaracetam (BRV) 2 (Experimental): 100 mg daily
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — 25 mg tablet - 50 mg daily for 17 weeks (or 21 weeks if down-titrated (50 mg > 20 mg) for subjects not participating in the follow-up study)
  Other Names: ucb 34714
  Arms: Brivaracetam (BRV) 1
Drug: Brivaracetam — 25 mg tablet - 100 mg daily for 17 weeks (or 21 weeks if down-titrated (100 mg > 50 mg > 20 mg) for subjects not participating in the follow-up study)
  Other Names: ucb 34714
  Arms: Brivaracetam (BRV) 2

SUMMARY:
Antiepileptic Drugs (AEDs) are the main treatment for epilepsy; however, only a limited number of AEDs are approved for use as monotherapy. The objective of this study is to evaluate the efficacy of BRV in the conversion of partial onset seizure patients from combination treatment to monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 16 to 75 years, both inclusive
* Well-characterized focal epilepsy or epileptic syndrome
* Subjects having at least 2 but not exceeding 40 partial onset seizures, whether or not secondarily generalized per 4 weeks during the 8-week Baseline Period
* Subjects on a stable dose of at least 1 but no more than 2 concomitant Antiepileptic Drugs (AEDs) with the second AED ≤ 50% of the minimum recommended maintenance dose

Exclusion Criteria:

* Seizure type IA non-motor as only seizure type
* History or presence of seizures occurring too frequently or indistinctly separated to be reliably counted during the 6 months preceding Visit 1 or during Baseline
* Other serious uncontrolled disease

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (68):
- United States (43):
  - Little Rock, Arkansas
  - Garden Grove, California
  - Loma Linda, California
  - Newport Beach, California
  - Riverside, California
  - Sacramento, California
  - Stanford, California
  - Denver, Colorado
  - Fort Collins, Colorado
  - Danbury, Connecticut
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Danville, Indiana
  - Elkhart, Indiana
  - Waldorf, Maryland
  - Grand Rapids, Michigan
  - Columbia, Missouri
  - Lebanon, New Hampshire
  - Albuquerque, New Mexico
  - Flushing, New York
  - Schenectady, New York
  - Charlotte, North Carolina
  - Oberlin, Ohio
  - Westerville, Ohio
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Jenkintown, Pennsylvania
  - Providence, Rhode Island
  - Austin, Texas
  - Bedford, Texas
  - San Antonio, Texas
  - Layton, Utah
  - Ogden, Utah
  - Burlington, Vermont
  - Bluefield, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Marshfield, Wisconsin
- France (4):
  - Béthune
  - Lille
  - Saint-Brieuc
  - Toulouse
- Germany (6):
  - Berlin
  - Bernau
  - Bielefeld
  - München
  - Münster
  - Ulm
- Hungary (4):
  - Budapest
  - Debrecen
  - Kecskemét
  - Szeged
- Italy (7):
  - Bergamo
  - Florence
  - Germaneto
  - Messina
  - Perugia
  - Pisa
  - Torino
- Spain (4):
  - Barcelona
  - Madrid
  - Murcia
  - Zaragoza

REFERENCES:
- [Result] Arnold S, Badalamenti V, Diaz A, Gasalla T, McShea C, Whitesides J, Fakhoury T. Conversion to brivaracetam monotherapy for the treatment of patients with focal seizures: Two double-blind, randomized, multicenter, historical control, Phase III studies. Epilepsy Res. 2018 Mar;141:73-82. doi: 10.1016/j.eplepsyres.2018.02.005. Epub 2018 Feb 12. PMID 29486396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-Center study started to enroll subjects in August 2008 and concluded in March 2010.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS). Subjects withdrawn due to meeting an exit criterion are included in the count of early discontinuations with a reason of "Adverse Event" or "Lack of efficacy" as reported by the Investigator.
Groups:
- Brivaracetam (BRV) 50 mg: 50 mg daily for 17 weeks (or 21 weeks if down-titrated (50 mg > 20 mg) for subjects not participating in the follow-up study).
- Brivaracetam (BRV) 100 mg: 100 mg daily for 17 weeks (or 21 weeks if down-titrated (100 mg > 50 mg > 20 mg) for subjects not participating in the follow-up study).
Period: Overall Study
Arm/Group | Brivaracetam (BRV) 50 mg | Brivaracetam (BRV) 100 mg
Started | 47 | 15
Completed | 14 | 7
Not Completed | 33 | 8
Not completed — Lack of Efficacy | 15 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Reason | 5 | 1
Not completed — SAE, non-fatal | 1 | 1
Not completed — AE, non-serious non-fatal | 8 | 1
Not completed — AE of unknown type | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intent-to-Treat Set (ITT), consisting of all randomized subjects with at least 1 intake of study medication.
Arm/Group | Brivaracetam (BRV) 50 mg | Brivaracetam (BRV) 100 mg | Total Title
Number analyzed (Participants) | 47 | 15 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 Years | 45 | 14 | 59
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.8) | 44.3 (15.9) | 40.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 11 | 38
  Male | 20 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Exit Rate at 112 Days After the Beginning of the Baseline Antiepileptic Drug (AED) Tapering Phase
Description: The cumulative exit rate was estimated using Kaplan-Meier methods and was based on the duration between start of the Evaluation Period (EP) and the earliest date the first exit criterion was met for each subject. Subjects completing the EP without meeting an exit criterion were censored on Day 112. The primary comparison was BRV 50 mg/day vs a historical control. The upper limit of the 2-sided 95 % Confidence Interval for the estimate was compared to the historical lower bound estimate of 0.722.
Time Frame: From Visit 4 (week 1) to the end of the Evaluation Period (week 17) (approximately 16 weeks)
Population: The Efficacy Analysis Set (EFF) consisted of all randomized subjects with at least 1 intake of study medication who also entered into the Baseline antiepileptic drug (AED) Tapering Phase (during the Evaluation Period) and started with the withdrawal of Baseline AEDs.
  The Outcome Measure was only pre-specified for the "Brivaracetam (BRV) 50 mg" Arm
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Efficacy Set (Brivaracetam 50 mg Treated Subjects): 50 mg daily for 17 weeks (or 21 weeks if down-titrated (50 mg > 20 mg) for subjects not participating in the follow-up study).
  The Efficacy Analysis Set (EFF) consisted of all randomized subjects with at least 1 intake of study medication who also entered into the Baseline antiepileptic drug (AED) Tapering Phase (during the Evaluation Period) and started with the withdrawal of Baseline AEDs.
Arm/Group | Efficacy Set (Brivaracetam 50 mg Treated Subjects)
Number analyzed (Participants) | 45
percentage of subjects | 0.474 [0.310 to 0.638]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Week 0 over the 1-week BRV Add-On Period and the 15-week Evaluation Period until the end fo Follow-Up Period (Week 23) or Early Discontinuation Visit.
Description: Adverse Events refer to the Intent-to-Treat (ITT) Set, consisting of all randomized subjects with at least 1 intake of study medication.
Arm/Group | Brivaracetam (BRV) 50 mg | Brivaracetam (BRV) 100 mg
Serious Adverse Events (participants affected / at risk) | 3/47 | 1/15
Other Adverse Events (participants affected / at risk) | 31/47 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (BRV) 50 mg (N=47) | Brivaracetam (BRV) 100 mg (N=15)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (4) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (BRV) 50 mg (N=47) | Brivaracetam (BRV) 100 mg (N=15)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2)
Irritability (General disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
White blood cells urine positive (Investigations) | 1 (1) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8) | 2 (2)
Convulsion (Nervous system disorders) | 5 (11) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 3 (4) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days